CLINICAL TRIAL: NCT07371455
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LWP779 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LWP779 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Longwood Pharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LW-A001
Record Dates: First submitted 2025-12-25; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single Ascending Dose - 150 mg (Experimental)
  Interventions: Drug: LWP779; Drug: Placebo of LWP779
- Single Ascending Dose - 300 mg (Experimental)
  Interventions: Drug: LWP779; Drug: Placebo of LWP779
- Single Ascending Dose - 600 mg (Experimental)
  Interventions: Drug: LWP779; Drug: Placebo of LWP779
- Single Ascending Dose - 900 mg (Experimental)
  Interventions: Drug: LWP779; Drug: Placebo of LWP779
- Single Ascending Dose - 1200 mg (Experimental)
  Interventions: Drug: LWP779; Drug: Placebo of LWP779

INTERVENTIONS:
Drug: LWP779 — Active
Drug: Placebo of LWP779 — Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial featuring both single ascending dose (SAD), food effect and multiple ascending dose (MAD) phases intended to evaluate the safety, tolerability, PK, PD, and active metabolites of LWP779 after oral administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent;
* 2. Males and females aged 18 to 65 years old (inclusive) at the time of signing the ICF.
* 3.No history of past or current diseases or abnormalities involving the cardiac, hepatic, renal, gastrointestinal, nervous, respiratory, or ocular systems, as well as psychiatric or metabolic abnormalities, that are clinically significant as judged by the investigator.
* 4.Participants must be confirmed healthy through medical history, VS, physical examination, clinical laboratory tests , and a 12-lead ECG;
* 5. Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and body weight not less than 50 kg at the time of screening and Day -1.
* 6. Participants must agree to take the investigator-approved effective contraceptive measures during the trial as required by the investigator.
* 7.Normal renal function (defined as eGFR ≥ 80 mL/min/1.73 m2) at screening and Day -1.
* 8. Ability to swallow and retain oral medication.
* 9.No suicidal ideation, as demonstrated by a score of "0" on the Columbia Suicide Severity Rating Scale (C-SSRS) at screening or Day -1.

Exclusion Criteria:

* 1.Known hypersensitivity to LWP779 or any of its constituents.
* 2.Known or suspected tumor.
* 3.History of unexplained syncope, symptomatic hypotension or hypoglycemia.
* 4.Presence of orthostatic hypotension at screening or Day -1.
* 5.Participants with any ocular diseases (e.g., glaucoma, fundus macular degeneration, corneal lesions, retinopathy, etc.).
* 6.Family history of long QTc syndrome; mean QTcF interval >450 msec for males and >470 msec for females or presence of any other mean ECG abnormality at screening or Day -1 deemed clinically significant by the PI/medical delegate.
* 7.Resting pulse rate <45 bpm or >100 bpm at screening, or Day -1.
* 8.Systolic blood pressure < 90 or >160 mm Hg and/or diastolic blood pressure < 50 or > 95 mm Hg at screening or Day -1.
* 9.History of unstable ischemic heart disease, recent (within 6 months of screening) myocardial infarction, or presence of clinically significant cardiac arrhythmia.
* 10.Ongoing liver disease or unexplained liver function test (LFT) elevations, defined as ALT, AST, gamma glutamyl transferase (GGT), alkaline phosphatase (ALP) or total/direct bilirubin > 1.5x ULN at screening or Day -1. Participants with confirmed Gilbert's syndrome will not be permitted to enroll in the study.
* 11.History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance deemed clinically significant by the PI/medical delegate.
* 12.History of cerebral hemorrhage (e.g., post-traffic accident), stroke, or cerebrovascular disease.
* 13.Participants judged by the PI/medical delegate to have any condition or history that may alter or increase bleeding tendency.
* 14.Participants regularly using drugs affecting coagulation function within 3 months before screening, or had received anticoagulant therapy such as heparin, low-molecular-weight heparin, fibrinolytic agents, etc. in the same timeframe.
* 15.Participants with conditions that may, in the opinion of the PI/medical delegate, significantly affect normal venous blood collection.
* 16.Positive results for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at screening.
* 17.Donated or lost >500 ml of blood in the previous 3 months prior to screening, donation of bone marrow or peripheral stem cells within 90 days prior to Day 1, or donation of plasma within 30 days prior to Day 1.
* 18.Participants who have participated in any investigational drug study within the past 3 months or 5 half-lives (whichever is longer) prior to dosing, or have participated in any investigational device study within the past 3 months prior to dosing.
* 19.Previous exposure to LWP779.
* 20.Use of prescription medications, vaccination, or any drugs known to induce or inhibit CYP3A4/5 or P-glycoprotein within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
* 21.Use of over-the-counter (OTC) medication or supplements (including vitamins, dietary supplements, herbal medicines, homoeopathy, etc.) within 14 days or 5 half-lives (whichever is longer), prior to receiving the first dose of study drug that might have impact on the clinical trial as per the PI/medical delegate's discretion. Acetaminophen (paracetamol) is permitted if provided maximum daily dose does not exceed 2000 mg.
* 22.Hospital admission or major surgery within 6 months prior to screening, or history of bariatric surgery.
* 23.A history of prescription drug misuse (as assessed by the PI/medical delegate), or positive urine drug screen at screening or Day -1.
* 24.Regular consumption of more than 10 standard alcoholic drinks per week or more than 4 standard alcoholic drinks on any one day, where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc/Vol], 100 mL wine [12% Alc/Vol], or 30 mL spirit [40% Alc/Vol]).
* 25.Consumes more than 2 cigarettes or equivalent nicotine-containing products per week, and/or is unwilling to abstain from the use of such products for 7 days prior to Day -1 through to EOS. Positive cotinine test at Day -1.
* 26.Use of cannabis or cannabidiol (CBD) containing products, in any form (e.g., edibles, oil, lotion, smoking) within 30 days prior to study drug administration on Day 1, regardless of legality within a given State, County or Region.
* 27.Participant is pregnant (as determined by pregnancy test result at screening or Day -1) or breastfeeding.
* 28.Participants who had consumed any food or beverage containing caffeine, alcohol, xanthine, Seville orange, pomelo, dragon fruit, starfruit, guava or grapefruit within 48 hours before each admission to the CRU.
* 29.A positive screen for alcohol at screening or Day -1.
* 30.Employee or family member of the Investigator (PI/medical delegate), study site personnel, or sponsor.
* 31.Food Effect study part only: unwilling to consume a high-fat meal consisting of eggs, bacon, butter, white bread and full cream milk.
* 32.Unable or unwilling to comply with the study restrictions and requirements
* 33.Participant developed an acute condition during the screening phase or before administration of the study drug; any other condition or finding that in the PI/medical delegate's opinion would put the participant or study conduct at risk if the participant were to be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of participants with a treatment-emergent adverse event (TEAE) | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD
12-lead electrocardiogram (ECG) (QT Interval) | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD
Number of participants with abnormal vital signs | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD
Number of participants with abnormal physical examination findings | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD
Columbia Suicide Severity Rating Scale (C-SSRS) | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD
  The Columbia Suicide Severity Rating Scale (C-SSRS) is used to assess suicidal ideation and suicidal behavior. Within the module "Answer for Actual Suicidal Attempts Only", the scoring range is 0 to 5. A score of 0 indicates no physical damage or very minor physical damage (e.g. surface scratches), and a score of 5 indicates death.
Number of participants with abnormal laboratory tests results | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD
Number of participants with abnormal ophthalmoscopic-examination findings | From baseline to Day 7 (±1) for SAD, baseline to Day16 (±2) for FE, baseline to Day 14 (± 2) for MAD

SECONDARY OUTCOMES:
C-QTc in the dose escalation part of SAD（in the dose groups of ≥300 mg） | Wthin 30 minutes before administration and to 24 hours after administration.
Maximum concentration (Cmax) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Time to reach Cmax (Tmax) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Total area under the concentration time curve (AUC) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Apparent terminal half-life (t1/2) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Terminal elimination rate constant (λz) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Apparent clearance (CL/F) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Apparent volume of distribution divided by bioavailability (Vd/F) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Lag time (tlag) of LWP779 and its active metabolites in plasma | Within 30 minutes before administration to 48 hours after single administration
Steady-state minimum concentration (Cmin,ss) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Steady-state maximum concentration (Cmax,ss) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Steady-state average concentration (Cavg,ss) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Area under the concentration-time curve from time zero to tau (AUC0-τ) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Time to reach Cmax (Tmax) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Terminal elimination rate constant (λz) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Apparent terminal half-life (t1/2) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Accumulation index (AUC0-τ (D7) / AUC0-τ (D1)) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.
Cmax (D7) / Cmax (D1)) of LWP779 and its active metabolites in plasma | Wthin 30 minutes before administration to 24 hours after multiple administration on Day 1 and Day 7, and 30 min pre-dose on Day 5 and Day 6.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Australia